CLINICAL TRIAL: NCT02670733
Title: Effect of Increased Positive End-expiratory Pressure on Intracranial Pressure in Different Respiratory Mechanic in Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Clinical Professor, Capital Medical University
Other Study IDs: K2015-023-01
Record Dates: First submitted 2016-01-26; First posted 2016-02-02 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-01

CONDITIONS: Acute Brain Injuries
Keywords: mechanical ventilation; positive end-expiratory pressure
MeSH Terms: conditions — Brain Injuries | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- high responsiveness of ICP to PEEP: After increasing positive end-expiratory pressure (PEEP) from 5 cmH2O to 15 cmH2O, intracranial pressure (ICP) increases above the median for the study population.
  Interventions: Procedure: Positive end-expiratory pressure
- low responsiveness of ICP to PEEP: After increasing positive end-expiratory pressure (PEEP) from 5 cmH2O to 15 cmH2O, the level of intracranial pressure (ICP) increases below the median for the study population.
  Interventions: Procedure: Positive end-expiratory pressure

INTERVENTIONS:
Procedure: Positive end-expiratory pressure — Positive end-expiratory pressure will be applied at 5 cmH2O and 15 cmH2O
  Other Names: PEEP

SUMMARY:
There are concerns that the use of positive end-expiratory pressure (PEEP) for the treatment of pulmonary complications in patients with brain injury may potentially elevate intracranial pressure (ICP), and deteriorate neurological status. It is suggested that both respiratory system compliance and ventricular compliance would contribute to the elevation of ICP when PEEP increases. In theory, PEEP may cause elevation of ICP by increasing intrathoracic pressure and diminish venous return. However, the transmission of PEEP into thoracic cavity depends on the properties of the lung and chest wall. Experimental study showed that when chest wall compliance is low, PEEP can significantly increases intrathoracic pressure; whereas low lung compliance can minimize airway pressure transmission. It is generally recognized that the lung compliance decreases in acute respiratory distress syndrome (ARDS) patients due to extensive alveolar collapse. However, it has been report that the elastance ratio (the ratio between elastance of the chest wall and the respiratory system, where elastance is the reciprocal of compliance) may vary from 0.2 to 0.8. Therefore, it is important to distinguish the compliance of the chest wall and the lung when investigating the effect of PEEP on ICP.

Because intrathoracic pressure (pleural pressure) is difficult to measure in clinical situations, esophageal pressure (Pes) is considered as a surrogate of intrathoracic pressure. In the present study, the investigators determine the effect of PEEP on intrathoracic pressure and ICP by Pes measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above;
2. Glasgow Coma Score ≤ 8;
3. Ventricular ICP monitor was placed for ICP monitoring and cerebrospinal fluid (CSF) drainage;
4. Need for mechanical ventilation with PEEP;
5. ARDS was diagnosed according to Berlin Definition.

Exclusion Criteria:

1. Hemodynamic instability requiring more than 10 μg/kg/min dopamine or more than 0.5 μg/kg/min norepinephrine;
2. ICP > 25 mmHg;
3. Esophageal varices;
4. History of esophageal or gastric surgery;
5. Evidence of active air leak from the lung, including bronchopleural fistula, pneumothorax, pneumomediastinum, or existing chest tube;
6. History of chronic obstructive pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe brain injured patients with ARDS
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in ICP level in different PEEP levels | Baseline ICP at PEEP of 5 cmH2O, and 15 minutes after increasing the PEEP level to 15 cmH2O

REFERENCES:
- [Derived] Chen H, Xu M, Yang YL, Chen K, Xu JQ, Zhang YR, Yu RG, Zhou JX. Effects of increased positive end-expiratory pressure on intracranial pressure in acute respiratory distress syndrome: a protocol of a prospective physiological study. BMJ Open. 2016 Nov 15;6(11):e012477. doi: 10.1136/bmjopen-2016-012477. PMID 27852713